CLINICAL TRIAL: NCT01803854
Title: CSP # 585 - Pilot Study: Gulf War Era Cohort and Biorepository
Brief Title: Gulf War Era Cohort and Biorepository
Acronym: CSP# 585
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 585; 11-09 (Other: Central IRB)
Record Dates: First submitted 2013-02-14; First posted 2013-03-04 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gulf War Era Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One EDTA tube of blood was collected from participants. All specimens have been processed and stored at the VA Central Biorepository (VACB) and its backup location for use in future research. One vial of buffy coat containing the DNA is stored. One aliquot of plasma was also extracted for storage from all samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gulf War Era Veterans: All Veterans who served in the uniformed services during 1990-1991 who signed consent forms, completed a survey, and provided a blood sample are included in the cohort.

SUMMARY:
The Gulf War Era Cohort and Biorepository pilot project collected epidemiological, survey, clinical, and environmental exposure data from Veterans who served during the 1990-1991 Gulf War Era. Approved researchers will be able to use these data and the blood samples to do future research about the health of Gulf War Era Veterans.

During the pilot, the recruitment response rate and processes were assessed. The results revealed several opportunities for improvement. For this reason, CSP 585 research activities transitioned to a qualitative phase to focus more on the Veteran voice. In this stage, research staff spoke with Gulf War Era Veterans through focus groups, interviews, and other activities such as events and meetings to learn more about Veterans' experiences and/or ideas on this and other Gulf War research projects. This phase provided new information that can help researchers create better recruitment processes for future projects involving Gulf War Era Veterans.

For more information on CSP 585, please contact Asia Johnson at asia.johnson4@va.gov and Christina Williams at christina.williams4@va.gov

DETAILED DESCRIPTION:
To date, the Department of Veterans Affairs (VA), the Department of Defense (DoD), and the Department of Health and Human Services have funded many research projects pertaining to the health consequences of military service in the 1990-1991 Gulf War. This past research represents a tremendous investment into understanding the medical conditions of these Veterans. However, many important questions remain to be answered about conditions affecting Gulf War Era Veterans. In addition, the Gulf War Era Veteran population is entering the age range at which the incidence of chronic diseases increases rapidly, and other questions are arising regarding the health and medical care of this important cohort.

The Gulf War Era Cohort and Biorepository pilot project collected epidemiological, survey, clinical, and environmental exposure data from Veterans who served during the 1990-1991 Gulf War Era. The goal was to enable the availability of blood specimens and health information for future immunologic, epidemiological, clinical, and health services research. During the pilot, the recruitment response rate and other operational and logistical aspects were assessed. Results indicated that our current recruitment processes were suboptimal for achieving our desired number of participants, and provide opportunities for improvement. To this end, CSP 585 research activities transitioned to a qualitative phase to focus more on the Veteran voice and learn more about how to effectively recruit Gulf War Era Veterans for a project like this. This phase provided new information that will inform recruitment processes for future projects involving Gulf War Era Veterans.

Specific Aims - The Gulf War Era Cohort and Biorepository pilot project was a minimal risk observational pilot project to test the processes needed to establish a research cohort and biorepository of Gulf War Era Veterans. There were no research questions or hypotheses. The pilot project had two specific aims:

1. assess the feasibility and efficacy of the planned recruitment, consenting, and blood drawing and shipping processes, and of modifications to the processes (if necessary); and
2. develop, test, and implement the database structures required for subject enrollment tracking, blood sample tracking, and data storage.

Veterans of the Gulf War Era were identified largely through existing VA and Department of Defense registries and databases. Some Veterans voluntarily joined and were eligible if they served in the military during 1990-91 without regard to actual deployment. The study database contains information collected from the Gulf War Era Veterans' Survey. Additional data will be collected from national VA and non-VA resources and from other studies of Gulf War Era Veterans.

Importance - There has been substantial research into the health care needs of Gulf War Era Veterans, but the incidence of chronic diseases that should be expected as this population ages is uncertain. Furthermore, the relationships between exposures, genetic susceptibility, and these illnesses have not been explored comprehensively in a large cohort. Data from the cohort described in this protocol includes survey data, plasma and access to VA and non-VA medical records, which can provide valuable resources for identifying risk factors as well as other chronic and aging related diseases. These data can then be used to identify the current and future health care needs of Gulf War Era Veterans to more effectively target programs towards them.

The intended users of the Gulf War Era Research Database and blood specimens are researchers who are specifically interested in illnesses affecting Gulf War Era Veterans, and researchers interested in the physical and mental health concerns that affect a population of this age group. The availability of a research cohort with the particular demographics and the documented experiences of Gulf War Era service will enable more detailed analyses regarding diagnosis and treatment of conditions affecting an aging population than is possible with administrative databases alone. With insights from analyses of data and blood specimens from this project, as well as others, the VA will be better able to focus interventions to improve diagnosis, treatment, and outcomes of care.

For more information on CSP 585, please contact Asia Johnson at asia.johnson4@va.gov and Christina Williams at christina.williams4@va.gov

ELIGIBILITY:
Inclusion Criteria:

* A potential participant must have been a member of the uniformed services during the 1990-1991 Gulf War era.
* A Veteran is eligible without regard to deployment or combat status and without regard to current or past user status in the Veterans Health Administration.

Exclusion Criteria:

* Veterans who did not serve in the military in 1990-1991 without regard to actual deployment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Veterans who served in the military in 1990-1991 without regard to actual deployment.
Sampling Method: Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2026-07-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Provenzale, MD MS, Study Chair — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khalil L, McNeil RB, Sims KJ, Felder KA, Hauser ER, Goldstein KM, Voils CI, Klimas NG, Brophy MT, Thomas CM, Whitley RL, Dursa EK, Helmer DA, Provenzale DT. The Gulf War Era Cohort and Biorepository: A Longitudinal Research Resource of Veterans of the 1990-1991 Gulf War Era. Am J Epidemiol. 2018 Nov 1;187(11):2279-2291. doi: 10.1093/aje/kwy147. PMID 30060060
- [Result] Brown MC, Sims KJ, Gifford EJ, Goldstein KM, Johnson MR, Williams CD, Provenzale D. Gender-based Differences among 1990-1991 Gulf War Era Veterans: Demographics, Lifestyle Behaviors, and Health Conditions. Womens Health Issues. 2019 Jun 25;29 Suppl 1(Suppl 1):S47-S55. doi: 10.1016/j.whi.2019.04.004. PMID 31253242
- [Result] Vahey J, Hauser ER, Sims KJ, Helmer DA, Provenzale D, Gifford EJ. Research tool for classifying Gulf War illness using survey responses: Lessons for writing replicable algorithms for symptom-based conditions. Life Sci. 2021 Oct 1;282:119808. doi: 10.1016/j.lfs.2021.119808. Epub 2021 Jul 6. PMID 34242657
- [Result] Gifford EJ, Vahey J, Hauser ER, Sims KJ, Efird JT, Dursa EK, Steele L, Helmer DA, Provenzale D. Gulf War illness in the Gulf War Era Cohort and Biorepository: The Kansas and Centers for Disease Control definitions. Life Sci. 2021 Aug 1;278:119454. doi: 10.1016/j.lfs.2021.119454. Epub 2021 Mar 31. PMID 33811897
- [Result] Vahey J, Gifford EJ, Sims KJ, Chesnut B, Boyle SH, Stafford C, Upchurch J, Stone A, Pyarajan S, Efird JT, Williams CD, Hauser ER. Gene-Toxicant Interactions in Gulf War Illness: Differential Effects of the PON1 Genotype. Brain Sci. 2021 Nov 25;11(12):1558. doi: 10.3390/brainsci11121558. PMID 34942860
- [Result] Gifford EJ, Boyle SH, Vahey J, Sims KJ, Efird JT, Chesnut B, Stafford C, Upchurch J, Williams CD, Helmer DA, Hauser ER. Health-Related Quality of Life by Gulf War Illness Case Status. Int J Environ Res Public Health. 2022 Apr 7;19(8):4425. doi: 10.3390/ijerph19084425. PMID 35457293
- [Result] Boyle SH, Upchurch J, Gifford EJ, Redding TS 4th, Hauser ER, Malhotra D, Press A, Sims KJ, Williams CD. Military exposures and Gulf War illness in veterans with and without posttraumatic stress disorder. J Trauma Stress. 2024 Feb;37(1):80-91. doi: 10.1002/jts.22994. Epub 2023 Nov 23. PMID 37997023
- [Result] Thompson AD Jr, Petry SE, Hauser ER, Boyle SH, Pathak GA, Upchurch J, Press A, Johnson MG, Sims KJ, Williams CD, Gifford EJ. Longitudinal Patterns of Multimorbidity in Gulf War Era Veterans With and Without Gulf War Illness. J Aging Health. 2025 Jun;37(5-6):281-291. doi: 10.1177/08982643241245163. Epub 2024 Apr 9. PMID 38591766
- [Result] Petry SE, Thompson AD Jr, Hauser ER, Lynch SM, Boyle SH, Upchurch J, Press A, Sims KJ, Williams CD, Gifford EJ. Characterizing Deficit Accumulation Among Gulf War Era Veterans. J Frailty Aging. 2024;13(3):300-306. doi: 10.14283/jfa.2024.44. PMID 39082776
- See also: An Assessment of Survey Measures Used Across Key Epidemiologic Studies of United States Gulf War I Era Veterans — http://www.ehjournal.net/content/pdf/1476-069X-12-4.pdf
- See also: Click here for more information about this study: CSP # 585 - Pilot Study: Gulf War Era Cohort and Biorepository — http://www.research.va.gov/programs/csp/585/default.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the pilot study (September 2014 through May 2016), recruitment materials were mailed to veterans from the stratified recruitment panel and those who self-nominated.The GWECB final enrollment included 1,275 "fully enrolled" veterans who completed all study requirements: 3 consenting documents, the GWECB survey, and a blood sample.
Period: Overall Study
Arm/Group | Gulf War Era Veterans
Started | 1275
Completed | 1275
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gulf War Era Veterans
Number analyzed (Participants) | 1275
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (8)
Age, Customized [Count of Participants; unit: Participants]
  Age group: ≤49 | 460
  Age group: 50-59 | 484
  Age group: 60-69 | 278
  Age group: ≥70 | 53
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 23 participants were missing sex data.
  Participants
    number analyzed (Participants) | 1252
    Female | 285
    Male | 967
Race/Ethnicity, Customized [Number; unit: participants] — The survey question pertaining to this characteristic allowed for more than one response (e.g., "check all that apply"); thus, numbers may not sum to participant totals.
  participants
    White | 922
    Black/African-American | 270
    American Indian/Alaska Native | 56
    Asian/Pacific Islander | 17
    Other Race | 45
    Missing Race Data | 32
    Not Spanish, Hispanic, or Latino | 1112
    Spanish, Hispanic, or Latino | 113
    Missing Ethnicity Data | 50

OUTCOME MEASURES:

1. Primary Outcome: VHA Health Care Utilization
Description: Use of VHA for health care in the past year
Time Frame: 20 months
Population: Twelve participants did not respond to the survey questions used to determine VHA user status.
Measure: Count of Participants; unit: Participants
Groups:
- VHA Health Care Utilization: Use of VHA for health care in the past year
Arm/Group | VHA Health Care Utilization
Number analyzed (Participants) | 1263
Participants
  Non-user | 679
  User | 584

2. Primary Outcome: Deployment
Description: Deployment in support of 1990-1991 Gulf War
Time Frame: 20 months
Population: Please note that the survey question pertaining to this characteristic allowed for more than one response (e.g., "check all that apply"); thus, the numbers sum to more than 1275 responses.
Measure: Number; unit: participants
Groups:
- Deployment Status: Self-reported deployment status during 1990-1991 Gulf War
Arm/Group | Deployment Status
Number analyzed (Participants) | 1275
participants
  Deployed to the Gulf | 900
  Did not deploy | 276
  Deployed elsewhere | 95
  Missing data | 21

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Gulf War Era Veterans
All-Cause Mortality (participants affected / at risk) | 0/1275
Serious Adverse Events (participants affected / at risk) | 0/1275
Other Adverse Events (participants affected / at risk) | 0/1275

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT01803854/Prot_SAP_ICF_000.pdf